CLINICAL TRIAL: NCT04597099
Title: Ability of Androgen-receptor Blockade to Normalize Progesterone-induced Augmentation of Gonadotropin Secretion in PCOS (CRM010)
Brief Title: Androgen Blockade and Progesterone Augmentation of Gonadotropin Secretion
Acronym: CRM010
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Chris McCartney, Professor of Medicine, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: HSR200016; R01HD102060 (NIH)
Record Dates: First submitted 2020-10-11; First posted 2020-10-22 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-11

CONDITIONS: PCOS; Polycystic Ovary Syndrome
Keywords: PCOS; Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Progesterone; Flutamide; Ortho Evra; Estradiol

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, double-blinded, crossover study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Flutamide (Experimental): Prior to the first or second admission (randomly determined), subjects will be pretreated for 4 weeks with Flutamide (250 mg twice daily)
  Interventions: Drug: Micronized progesterone; Drug: Flutamide; Drug: Estradiol patch
- Placebo (Placebo Comparator): Prior to the first or the second admission (randomly determined), participants will be pretreated for 2 weeks with placebo (twice daily).
  Interventions: Drug: Micronized progesterone; Drug: Placebo; Drug: Estradiol patch

INTERVENTIONS:
Drug: Micronized progesterone — oral micronized progesterone suspension, 100 mg oral dose at 0800 during each study admission
  Other Names: progesterone
Drug: Placebo — Placebo contains only inert ingredients and is not expected to exert any direct physiological effects.
  Arms: Placebo
Drug: Flutamide — Flutamide, 250 mg taken orally twice daily for four weeks before study admission.
  Arms: Flutamide
Drug: Estradiol patch — Two 0.1 mg/day transdermal estradiol patches will be applied 3 days prior to each inpatient admission; on the morning of study admission, these two patches will be removed and immediately replaced with two new 0.1 mg/day patches.
  Other Names: Vivelle

SUMMARY:
This study is trying to find out if flutamide (a medication that blocks the effects of testosterone) may help normalize an aspect of pituitary function (specifically, gonadotropin surge generation) in PCOS. This is a randomized, placebo-controlled, double-blinded, crossover study. The investigators hypothesize that in estradiol-pretreated women with PCOS, acute progesterone augmentation of FSH release (positive feedback) will be enhanced by flutamide.

DETAILED DESCRIPTION:
Women with PCOS appear to exhibit impaired progesterone (P4) augmentation of gonadotropin release (positive feedback), and this is at least partly independent of BMI differences. To test more directly the role of hyperandrogenemia/hyperandrogenism (HA), we will assess if the androgen-receptor blocker flutamide enhances P4 augmentation of gonadotropin release in estradiol (E2)-treated women with PCOS. We will study 10 women with PCOS. This is a randomized, placebo-controlled, double-blinded, crossover study, with subjects undergoing two assessments of P4 positive feedback - once after 4 weeks' pretreatment with flutamide and once after 4-weeks' pretreatment with placebo (in random order). We will assess P4 positive feedback via frequent sampling for 16 hours. Subjects will be pretreated for 3 days (prior to CRU admission) with transdermal E2 (0.2 mg/day), starting no earlier than cycle day 7. Subjects will be admitted to the CRU the evening of day 3 of E2 treatment. Starting at 0200 h, blood will be collected for 16 hours. After 6 h of sampling (0800 h), subjects will receive a single oral dose of P4. A second CRU admission - performed at least 2 months later to permit adequate washout of flutamide (as needed) - will be identical to the first except that placebo pretreatment will be exchanged for flutamide pretreatment or vice versa. We will assess the P4-mediated augmentation of FSH release, with secondary endpoints including the P4-mediated augmentation of LH release. We hypothesize that in E2-pretreated women with PCOS, acute P4 augmentation of FSH release (positive feedback) will be enhanced by androgen-receptor blockade (flutamide).

ELIGIBILITY:
Inclusion Criteria:

* Post-pubertal (> 4 years post-menarche) adult woman aged 18-30 years
* PCOS, defined as clinical and/or laboratory evidence of hyperandrogenism (hirsutism and/or elevated serum [calculated] free testosterone concentration) plus ovulatory dysfunction (irregular menses, fewer than 9 per year), but without evidence for other potential causes of hyperandrogenism and/or ovulatory dysfunction
* General good health (excepting overweight, obesity, hyperandrogenism, PCOS, and adequately-treated hypothyroidism)
* Capable of and willing to provide informed consent
* Willing to strictly avoid pregnancy with use of reliable non-hormonal methods during the study period

Exclusion Criteria:

* Inability/incapacity to provide informed consent
* Males will be excluded (PCOS is unique to females)
* Age < 18 years or > 30 years (ovarian reserve may decrease beyond age 30)
* Obesity resulting from a well-defined endocrinopathy or genetic syndrome
* Positive pregnancy test or current lactation
* Evidence for non-physiologic or non-PCOS causes of hyperandrogenism and/or anovulation
* Evidence of virilization (e.g., rapidly progressive hirsutism, deepening of the voice, clitoromegaly)
* Total testosterone > 150 ng/dl, which suggests the possibility of virilizing ovarian or adrenal tumor
* DHEA-S elevation > 1.5 times the upper reference range limit. Mild elevations may be seen in PCOS, and will be accepted in these groups
* Early morning 17-hydroxyprogesterone > 200 ng/dl measured in the follicular phase, which suggests the possibility of congenital adrenal hyperplasia (if elevated during the luteal phase, the 17-hydroxyprogesterone will be repeated during the follicular phase). NOTE: If a 17-hydroxyprogesterone > 200 ng/dl is confirmed on repeat testing, an ACTH stimulated 17-hydroxyprogesterone < 1000 ng/dl performed by the subject's personal physician will be required for study participation.
* Abnormal thyroid stimulating hormone (TSH): Note that subjects with stable and adequately treated primary hypothyroidism, reflected by normal TSH values, will not be excluded.
* Hyperprolactinemia > 20% higher than the upper limit of normal. Mild prolactin elevations may be seen in women with PCOS, and elevations within 20% higher than the upper limit of normal will be accepted in this group.
* History and/or physical exam findings suggestive of Cushing's syndrome, adrenal insufficiency, or acromegaly
* History and/or physical exam findings suggestive of hypogonadotropic hypogonadism (e.g., symptoms of estrogen deficiency) including functional hypothalamic amenorrhea (which may be suggested by a constellation of symptoms including restrictive eating patterns, excessive exercise, psychological stress, etc.)
* Persistent hematocrit < 37% and hemoglobin < 12 g/dl
* Severe thrombocytopenia (platelets < 50,000 cells/microliter) or leukopenia (total white blood count < 4,000 cells/microliter)
* Previous diagnosis of diabetes, fasting glucose > or = 126 mg/dl, or a hemoglobin A1c > or = 6.5%
* Given that this study involves flutamide use, any liver panel abnormality will be grounds for exclusion
* Significant history of cardiac or pulmonary dysfunction (e.g., known or suspected congestive heart failure, asthma requiring intermittent systemic corticosteroids, etc.)
* Decreased renal function evidenced by GFR < 60 ml/min/1.73m2
* A personal history of breast, ovarian, or endometrial cancer
* History of allergy to micronized progesterone, flutamide, or transdermal estradiol
* BMI < 18 or > 40 kg/m2
* Due to the amount of blood being drawn, volunteers with body weight < 110 pounds must be excluded

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This is a study regarding PCOS, so only females will be eligible
Enrollment: 10 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in mean FSH concentration with progesterone administration | After 4 weeks of placebo administration
  Change in mean FSH concentrations (post-progesterone FSH concentrations vs. pre-progesterone FSH concentrations)
Change in mean FSH concentration with progesterone administration | After 4 weeks of flutamide administration
  Change in mean FSH concentrations (post-progesterone FSH concentrations vs. pre-progesterone FSH concentrations)

SECONDARY OUTCOMES:
Change in mean LH concentration with progesterone administration | After 4 weeks of placebo administration
  Change in mean LH concentrations (post-progesterone LH concentrations vs. pre-progesterone LH concentrations)
Change in mean LH concentration with progesterone administration | After 4 weeks of flutamide administration
  Change in mean LH concentrations (post-progesterone LH concentrations vs. pre-progesterone LH concentrations)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M McCartney, MD, Principal Investigator — Univsersity of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No